CLINICAL TRIAL: NCT05363033
Title: Evaluation of a Sarcopenia Prediction Model and Development and Effectiveness of a Nursing Guidance Mobile App
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Pei-Hung Liao, Assistant Professor, National Taipei University of Nursing and Health Sciences
Other Study IDs: 108A-06
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Prediction of High-risk Populations for Sarcopenia
Keywords: artificial intelligence, nursing, nursing guidance mobile application, prediction model, sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group: Using a one-group pretest-posttest design
  Interventions: Device: sarcopenia nursing guidance mobile application was developed

INTERVENTIONS:
Device: sarcopenia nursing guidance mobile application was developed — The application enhanced participants' sarcopenia-related knowledge and awareness regarding self-care

SUMMARY:
We evaluated a model for the prediction of high-risk populations for sarcopenia in home settings, developed a sarcopenia nursing guidance mobile application, and assessed the effectiveness of this application in influencing sarcopenia-related knowledge and self-care behavior among participants.

ELIGIBILITY:
Inclusion criteria were being a member of the public, aged ≥20 years and <80 years, and having experience using mobile devices or smartphones. Exclusion criteria were not belonging to a high-risk population for sarcopenia and/or being unable to use the application platform.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We adopted the convenient sampling method to recruit 120 participants-those who visited the hospital regularly and their accompanying family members
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
changes in sarcopenia-related knowledge and awareness regarding self-care | 2019~2022
  In this study, the mobile app significantly improved sarcopenia-related knowledge and awareness regarding self-care among the participants

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Hsin General Hospital, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liao PH, Huang YJ, Ho CS, Chu W. Application of machine learning and its effects on the development of a nursing guidance mobile app for sarcopenia. BMC Nurs. 2023 Oct 9;22(1):369. doi: 10.1186/s12912-023-01545-w. PMID 37814285